CLINICAL TRIAL: NCT02952066
Title: Expressions of TRPV1 in Airway of Asthmatics
Acronym: TRPV1
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Prior to any participant enrollment, the PI opted to not move forward with the study.
Sponsor: Lu Yuan Lee (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor-Investigator, Lu Yuan Lee, Sponsor/PI, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 15-0349-F6A; U01AI123832 (NIH)
Record Dates: First submitted 2016-10-29; First posted 2016-11-02 (Estimated); Last update posted 2021-06-14 (Actual); Status verified 2021-06

CONDITIONS: Moderate Persistent Asthma; Severe Persistent Asthma; Nodule Solitary Pulmonary; Pulmonary Atelectasis
MeSH Terms: conditions — Solitary Pulmonary Nodule; Pulmonary Atelectasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TRP1 Density (Experimental): Bronchial Biopsy: During the biopsy procedure the investigator will collect five bronchial specimens (1-2 cubic millimeters) each the major, lobar and segmental bronchi.
  Interventions: Procedure: Bronchial biopsy

INTERVENTIONS:
Procedure: Bronchial biopsy — Bronchial tissue taken during biopsy

SUMMARY:
The purpose of this study is to measure the density of a temperature-sensitive protein, named TRPV1, in the airway mucosa tissue of both non-asthmatic and moderate to severe persistent asthmatic patients. This study may generate information for developing new therapeutic strategy.

DETAILED DESCRIPTION:
The research procedure will be conducted at University of Kentucky A.B. Chandler Hospital dedicated bronchoscopy suite located on third floor of Pavilion H module room #2, and will be performed only once as part of a standard of care bronchoscopy procedure scheduled by the participants pulmonary physician. This entire study (biopsy) will add 10 minutes or less. Following the biopsy, and after being discharged from the hospital, the participant's study participation will end.

Bronchial Biopsy: The investigator will collect five lung (bronchial) specimens (1-2 cubic millimeters each) from three zones of the participant's airway which will be individually coded, and stored for the computer image analysis of TRPV1 in the investigator's laboratory. Following analysis the samples will be destroyed. The results of the analysis cannot be used for determining a clinical diagnosis. Therefore, the investigator will not provide any findings to either the participant or their physician.

Participants will not get any personal benefit from taking part in this study. Their willingness to take part in this research study, may, in the future help doctors better understand and/or treat patients with asthma.

There will be no cost to the participant for having the bronchial biopsy performed.

Participants will not receive any rewards or payment for taking part in the study.

ELIGIBILITY:
Inclusion Criteria:

* Competent to understand informed consent
* Diagnosis of moderate to severe persistent allergic asthma.
* Clinical need for diagnostic bronchoscopy for assessment of asthmatic symptoms (e.g., to assess presence of chronic infection with non-tuberculous mycobacteria or other infectious agents as a cause for lack of asthma control) or therapeutic bronchoscopy for management of asthmatic symptoms (e.g., thermoplasty).
* Asthmatic subjects with history of positive skin test to confirm presence of allergy.
* Asthmatic subjects with pre-albuterol forced expiratory volume in the first second (FEV1) of <70% of the predicted value.
* Non-asthmatic patients will include those patients with solitary pulmonary nodules and healthy individuals with acute lung atelectasis (e.g. airway blocked by mucus plugs or foreign object).
* Scheduled for a diagnostic or therapeutic bronchoscopy procedure.

Exclusion Criteria:

* Inability to perform pulmonary function testing
* Unstable asthma control for asthmatic subjects
* An asthma exacerbation within the past month
* History of intubation for asthma
* History of smoking
* History of prematurity
* History of any lung disease or disorder except asthma
* History of congenital or acquired heart disease
* Pregnant/lactating females
* Any serious concurrent systemic disease including but not limited to diabetes, coronary artery disease, vasculitis, etc.
* History of heart arrhythmias including supraventricular tachycardia

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2017-09-20 (Actual); Primary Completion 2018-11-20 (Actual); Study Completion 2018-11-20 (Actual)

PRIMARY OUTCOMES:
TRPV1 density in airway mucosa tissue | one year

CONTACTS AND LOCATIONS:
Overall Officials: Lu-Yan Lee, PhD, Study Chair — University of Kentucky; Mehdi Khosravi, MD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky Medical Center, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No